CLINICAL TRIAL: NCT04891003
Title: The Identification of Optimal Ultrasonografic Tecniques for Determining the Location , Size and the Surgical Methods of Intestinal Endometriotric Nodules
Acronym: Sonography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Resul Karakuş, Specialist, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: 2020/147
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: ULTRASONOGRAPHY; Endometriosis, Rectum
Keywords: Endometriosis; Diagnostic Imaging
MeSH Terms: conditions — Endometriosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients Diagnosed with Endometriosis (or endometrioma alone): Nulliparous patients who had diagnosed with endometriosis, no additional gynecological patology such as myoma uteri, polype, a history of pelvic inflammatuar disease, a history of cervical or uterine surgery, uterine anomalies
  Interventions: Diagnostic Test: Ultrasonography
- Patients With No Gynecological Pathology: Nulliparous patients who had not diagnosed with endometriosis, no additional gynecological patology such as myoma uteri, polype, a history of pelvic inflammatuar disease, a history of cervical or uterine surgery, uterine anomalies
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — The identification of optimal ultrasonografic tecniques for determining the location , size and the surgical methods of intestinal endometriotric nodules.

SUMMARY:
The identification of optimal ultrasonografic tecniques for determining the location , size and the surgical methods of intestinal endometriotric nodules

DETAILED DESCRIPTION:
Nulliparous patients who had diagnosed with endometriosis ( endometrioma and/or deep endometriosis) without additional gynecological patology applying for routine gynecological check-up to Zeynep Kamil Training and Research Hospital, Gnecology and Obstetrics Clinic between March 2020 and March 2021 will be included in the study.Inclusion criteria in the study. Inclusion criterias are the presence of endometrioma and/or endometriosis diagnosed with ultrasonographic evaluation, nulliparity,no additional gynecological patology such as myoma uteri, polype, a history of pelvic inflammatuar disease, a history of cervical or uterine surgery, uterine anomalies as well as patients in the control group will be nulliparous and have no gynecological patology including endometrioma and/or endometriosis.All patients will be evaluated in the follicular phase.With the ultrasonographic examination, the uterine version ( anteversion or retroversion) will be evaluated, the length of the uterus (from fundus to cervix on the saggital axis), the anterior-posterior widest uterin length ( at the level of corpus uteri), the cervical length (the distance between the internal os and external os), the cervical anteroposterior length ath the internal os level and the servical canal length at the internal os level, uterocervical angle (the angle between the longitudinal axis of the cervix and the longitudinal axis of the uterine body will be measured three times consecutively , the avarage of the three measurements will be recoreded).with the 90 degree rotation of the probe at the transverse axis the width of the widest corpus level of uterus and the width of the cervix will be measured.Measurements will be made by the same clinician with the same ultrasound device. These measurements and the patients' age, BMI(body mass index), menarche cycle duration, dysmenorrhea, dyspareunia, family history in terms of endometriosis, endometrisosis stage will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with deep infiltrative endometriosis and intestinal involvement
* Treatment will be done surgically
* Patients should be nonvirgin

Exclusion Criteria:

* Patient has one or more extra -intestinal findings of deep infiltrative endometiosis

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — 18-45
Study Population: Non- virgin Female Patients having only intestinal findings of deep infiltrative endometriosis aged between 18-45 years old ,
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-05-08 (Estimated)

PRIMARY OUTCOMES:
Endometriosis,intestinal | 4 months
  Ultrrasonographic imaging of endometriosis

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Childrens Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)